CLINICAL TRIAL: NCT05925192
Title: Profile of Chronic Musculoskeletal Pain Patients Related to Treatment Adherence and Virtual Reality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Torres Sánchez, PT, PhD, Principal investigator, Universidad de Granada
Other Study IDs: DMCRV-01
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Chronic Musculoskeletal Pain
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic musculoskeletal pain patients: Chronic musculoskeletal pain patients
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — N/A - observational study

SUMMARY:
Lack of adherence is one of the main problems of chronic musculoskeletal pain treatment. To improve adherence it is essential to take into account the characteristics of the patients and their thoughts and beliefs about pain. Virtual reality can present some advantages in the face of these problems too.

The objective of this study is to evaluate the profile of chronic musculoskeletal pain patients, the barriers associated with lack of adherence to treatment, and the interest of virtual reality in rehabilitation.

DETAILED DESCRIPTION:
* Background: Lack of adherence is one of the main problems of chronic musculoskeletal pain treatment. To improve adherence it is essential to take into account the characteristics of the patients and their thoughts and beliefs about pain. Virtual reality can present some advantages in the face of these problems too.
* Objectives: Evaluate the profile of chronic musculoskeletal pain patients, the barriers associated with lack of adherence to treatment, and the interest of virtual reality in rehabilitation.
* Methodology: Observational study. The profile of chronic musculoskeletal pain patients will be described. Patients will be recruited using the snowball method. The evaluation will be carried out via telematics through the use of videoconference and surveys. We will evaluate chronic pain and characteristics, kinesiophobia, functionality, quality of life, psychosocial aspects and other related outcomes. We will identify barriers associated to treatment adherence and we will evaluate patients' perception of rehabilitation with virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain (≥ 3 months)
* Adults (≥ 18 years)
* Have a computer or mobile device/Basic knowledge and access to the internet
* Wish to participate in the study and sign the informed consent

Exclusion Criteria:

All those participants who present any physical pathology or of any kind that imply an inability to understand the necessary instructions to carry out the study will be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic musculoskeletal pain patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline
  To assess pain intensity using the verbal numeric pain scale. Scores range from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate greater intensity.
Pain Intensity and chronic pain interference | Baseline
  To assess pain intensity and chronic pain interference using the graded chronic pain scale. Scores range from 0 (no pain/no interference) to 10 (worst pain imaginable/unable to carry on any activities). Higher scores indicate greater intensity or interference.
Pain Severity | Baseline
  To assess pain severity using the brief pain inventory. Scores range from 0 (no pain/does not interfere) to 10 (worst pain imaginable/completely interferes). Higher scores indicate greater severity.
Awareness, Consciousness, Vigilance and Observation of pain | Baseline
  To assess awareness, consciousness, vigilance and observation of pain using the pain vigilance and awareness questionnaire. Scores range from 0 (never) to 5 (always). The total questionnaire scores range between 0 and 80. Higher scores indicate greater awareness, consciousness, vigilance and observation of pain.
Chronic Pain Acceptance | Baseline
  To assess chronic pain acceptance using the chronic pain acceptance questionnaire. Scores range from 0 (never true) to 6 (it is always true). Higher scores indicate greater acceptance.
Neurophysiology of Pain | Baseline
  To assess neurophysiology of pain using the neurophysiology of pain questionnaire. Scores range from 0 to 13 (sum of all correct items).

SECONDARY OUTCOMES:
Kinesiophobia | Baseline
  To assess kinesiophobia using the TAMPA scale of kinesiophobia. Scores range from 1 (totally disagree) to 4 (totally agree). The final score can range between 11 and 44 points, with higher scores indicating greater perceived kinesiophobia.
Catastrophizing of pain | Baseline
  To assess catastrophizing of pain using the pain catastrophizing scale. Scores range from 0 (nothing at all) to 4 (all the time). The final score range between 0 and 52 points, with higher scores indicating greater levels of catastrophism.
Functionality | Baseline
  To assess functionality using the functional independence measure. Scores range from 1 (total assistance) to 7 (complete independence). The final score range between 18 and 126 points, with higher scores indicating greater independence.
Disability | Baseline
  To assess disability using the world health organisation disability assessment. . Scores range from 1 (none) to 5 (extreme). The final score range between 12 and 60 points, with higher scores indicating worst disability.
Level of movement related to space | Baseline
  To assess level of movement related to space using the life space questionnaire. Scoring is based on "yes" (1 point) or "no" (2 points) answers. The more answers that do "no" exist in the questionnaire, the lower their level of movement in the space will be.
Health-related Quality of Life | Baseline
  To assess health-related quality of life using the euroqol-5d. Total score range from 1 (best health status) to 0 (death). The second part of the euroqol-5d is visual analogue scale that goes from 0 (worst state of health imaginable) to 100 (best state of health imaginable).
Sleep Quality | Baseline
  To assess sleep quality using the Pittsburgh sleep quality index. The overall score ranges from 0 to 21 points. "0" indicates ease of sleeping and "21" severe difficulty in all areas.
Depression and anxiety | Baseline
  To assess depression and anxiety using the hospital anxiety and depression scale. The total score ranges from 0 to 21 on each subscale, where a higher score is indicative of more severe symptoms.
Physical activity | Baseline
  To assess physical activity using the international physical activity questionnaire. This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in Metabolic Equivalent (MET)-min/week and time spent sitting.
Work performance | Baseline
  To assess work performance using the work role functioning questionnaire. Total score range from 0% (difficulty all the time) to 100 % (no difficulty at any time).
Social support | Baseline
  To assess social support using the medical outcomes study social support survey
Treatment information and barriers associated to treatment adherence | Baseline
  To assess information about treatment and barriers associated to treatment adherence using Likert-type questions range from 1 (totally disagree) to 5 (totally agree).
Barriers associated to doing exercise therapy | Baseline
  To assess barriers associated to doing exercise therapy using the exercise therapy burden questionnaire. Scores range from 0 (totally disagree) to 10 (totally agree).
Patients' perception to virtual reality rehabilitation | Baseline
  To assess patients' perception to virtual reality rehabilitation using Likert-type questions and yes or no questions

CONTACTS AND LOCATIONS:
Overall Officials: Irene Torres Sánchez, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain